CLINICAL TRIAL: NCT01734928
Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Compare the Efficacy and Safety of Pomalidomide, Bortezomib and Low-Dose Dexamethasone Versus Bortezomib and Low-Dose Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Safety and Efficacy of Pomalidomide, Bortezomib and Low-dose Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Acronym: OPTIMISMM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-007
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Pomalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pomalidomide, Bortezomib and Low Dose Dexamethasone (Experimental): 4 mg of Pomalidomide will be taken orally on Days 1-14 of a 21-day cycle along with 1.3 mg/m2 of Bortezomib administered subcutaneously on Days 1, 4, 8 and 11 of 21 days for cycles 1 -8 and on days 1, 8 of 21 days for cycle 9 and onward until disease progression, and Dexamethasone 20 mg/day [≤ 75 years old] or 10 mg/day [> 75 years old] orally on days 1, 2, 4, 5, 8, 9, 11, 12 of 21 days for cycles 1-8 and on days 1, 2,8, 9 of 21 days for cycles 9 and onward until disease progression.
  Interventions: Drug: Pomalidomide; Drug: Bortezomib; Drug: Dexamethasone
- Bortezomib and Low Dose Dexamethasone (Active Comparator): 1.3 mg/m2 of Bortezomib will be administered subcutaneously on Days 1, 4, 8 and 11 of 21 days for cycles 1 -8 and on Days 1, 8 of 21 days for cycle 9 and onward until disease progression along with Dexamethasone 20 mg/day [≤ 75 years old]or 10 mg/day [> 75 years old] orally on days 1, 2, 4, 5, 8, 9, 11, 12 of 21 days for cycles 1-8 and on Days 1, 2, 8, 9 of 21 days for cycles 9 and onward until disease progression.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — Pomalidomide 4 mg will be taken orally on Days 1-14 of a 21-day cycle.
  Other Names: Oral Pomalidomide; CC-4047
  Arms: Pomalidomide, Bortezomib and Low Dose Dexamethasone
Drug: Bortezomib — Bortezomib 1.3 mg/m2 will be administered subcutaneously on Days 1, 4, 8 and 11 of 21 days for cycles 1 -8 and on Days 1, 8 of 21 days for cycle 9 and onward until disease progression.
  Other Names: Velcade
Drug: Dexamethasone — Dexamethasone 20 mg/day [≤ 75 years old] or 10 mg/day [>75 years old] will be taken orally on Days 1, 2, 4, 5, 8, 9, 11, 12 of 21 days for cycles 1-8 and on Days 1, 2, 8, 9 of 21 days for cycles 9 and onward until disease progression.

SUMMARY:
The purpose of this study is to compare the efficacy of the combination of pomalidomide, bortezomib and low dose dexamethasone to the combination of bortezomib and low dose dexamethasone in participants with relapsed/refractory multiple myeloma. This study will also assess how safe the combination of pomalidomide, bortezomib and low dose dexamethasone is compared to the combination of bortezomib and low dose dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years at the time of signing informed consent.
* Must have documented diagnosis of multiple myeloma and have measureable disease by serum and urine protein electrophoresis.
* Must have had at least 1 but no greater than 3 prior anti-myeloma regimens.
* Must have documented disease progression during or after their last anti-myeloma therapy.
* All subjects must have received prior treatment with a lenalidomide containing regimen for at least 2 consecutive cycles.

Exclusion Criteria:

* Documented progressive disease during therapy or within 60 days of the last dose of a bortezomib-containing therapy under the 1.3 mg/m^2 dose twice weekly dosing schedule.
* Peripheral neuropathy Grade 3, Grade 4 or Grade 2 with pain within 14 days prior to randomization.
* Non-secretory multiple myeloma.
* Subjects with severe renal impairment requiring dialysis.
* Previous therapy with pomalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers-Squibb, Study Director — Bristol-Myers Squibb; Amine Bensmaine, MD, Study Director — Celgene Corporation
Locations (321):
- United States (92):
  - Southern Cancer Center, Mobile, Alabama
  - Arizona Oncology, Tucson, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - University of California San Francisco Fresno Campus, Fresno, California
  - Marin Oncology Associates, Greenbrae, California
  - Moore UCSD Cancer Center, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Local Institution - 153, Southington, Connecticut
  - George Washington Medical Center, Washington D.C., District of Columbia
  - Lynn Cancer Institute, Boca Raton, Florida
  - University Cancer Institute, Boynton Beach, Florida
  - Broward Oncology Associates PA, Fort Lauderdale, Florida
  - Broward Oncology Assoc., Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Alves Domenech Oncology and Hematology Clinic, Hollywood, Florida
  - Palm Beach Cancer Institute, LLC, West Palm Beach, Florida
  - Local Institution - 135, Marietta, Georgia
  - Northwest Georgia Oncology Centers, PCWilliam S. Gibbons Center Research Institute, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Western Kentucky Hematology and Oncology Group, PSC, Paducah, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - Cancer Care of Maine, Bangor, Maine
  - Local Institution - 132, Bangor, Maine
  - St. Agnes - Medical Center, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Local Institution - 125, Bethesda, Maryland
  - Medstar Health Research Institute, Hyattsville, Maryland
  - Local Institution - 299, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 100, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Local Institution - 298, Boston, Massachusetts
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Local Institution - 178, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Detroit Clinical Research Center, Lansing, Michigan
  - Beaumont Cancer Center, Royal Oak, Michigan
  - Essentia Health Duluth CCOP, Duluth, Minnesota
  - Metro MN CCOP, Saint Louis Park, Minnesota
  - Columbia Comprehensive, Jefferson City, Missouri
  - Kansas City VA Medical Center University of Kansas Medical Center, Kansas City, Missouri
  - St. John's Clinic Cancerand Hematology - Springfield, Springfield, Missouri
  - St John's Mercy Medical Center, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - CarePoint Health Research Institute, Jersey City, New Jersey
  - Hematology-Oncology Associates of NNJ, P, Morristown, New Jersey
  - Somerset Hematology-Oncology Associates, Somerville, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Local Institution - 186, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Eastern Institute of Medical Sciences, Greenville, North Carolina
  - Boice-Willis Clinic P.A., Rocky Mount, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Local Institution - 111, Canton, Ohio
  - MetroHealth Medical Systems, Cleveland, Ohio
  - Mid Ohio Oncology Hematology Inc, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Med Univ of South Carolina, Charleston, South Carolina
  - Spartanburg Regional Healthcare System - Gibbs Cancer Center & Research Institute, Spartanburg, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Local Institution - 167, Watertown, South Dakota
  - Prairie Lakes Health Care System, Watertown, South Dakota
  - University of Tennessee Medical Center - Cancer Institute, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Local Institution - 114, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center Francis Street Medical Center, Fort Sam Houston, Texas
  - Local Institution - 103, Fort Sam Houston, Texas
  - Local Institution - 130, Houston, Texas
  - Northwest Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Utah Cancer Specialist, Salt Lake City, Utah
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
  - Swedish Cancer Inst, Seattle, Washington
  - Medical Oncology Associates, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Local Institution - 139, Morgantown, West Virginia
  - West Virginia University CTRU, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Local Institution - 136, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Austria (6):
  - Hospital St. Polten, Sankt Pölten
  - Local Institution - 523, Sankt Pölten
  - Local Institution - 480, Vienna
  - Medical University of Vienna, Vienna
  - Local Institution - 481, Vienna
  - Wilhelminenspital-Center for Hematology and Oncology, Vienna
- Canada (9):
  - Local Institution - 308, Oshawa, Ontario
  - RSM Durham Regional Cancer Center - Lakeridge Health Oshawa, Oshawa, Ontario
  - CSSS Champlain Charles LeMoyne, Greenfield Park, Quebec
  - Local Institution - 301, Greenfield Park, Quebec
  - Centre De Sante Et De Services Sociaux De Rimouski-Neigette, Rimouski, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Hospital Fleurimont, Sherbrooke, Quebec
  - Local Institution - 307, Sherbrooke, Quebec
  - Local Institution - 304, Halifax
  - Queen Elizabeth II Health Sciences Centre, Halifax
- Denmark (8):
  - Aarhus University Hospital, Aarhus
  - Local Institution - 447, Aarhus
  - Copenhagen University Hospital Rigshosptalet, Copenhagen
  - Local Institution - 506, Copenhagen
  - Local Institution - 400, Odense
  - Odense University Hospital, Odense
  - Local Institution - 499, Vejle
  - Vejle Hospital, Vejle
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Local Institution - 455, Helsinki
  - Hyvinkaa Hospital, Hyvinkää
  - Local Institution - 510, Hyvinkää
- France (21):
  - Centre Hospitalier de la cote basque, Bayonne
  - Local Institution - 469, Bayonne
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Local Institution - 498, Chalon-sur-Saône
  - CHU Hotel, Grenoble
  - Local Institution - 483, Grenoble
  - GH Institut Catholique St Vincent, Lille
  - CHRU de Lille-Hopital Claude Huriez, Lille
  - Local Institution - 476, Lille
  - CHRU Hotel Dieu, Nantes
  - Local Institution - 486, Nantes
  - Groupement Hospitalier Universitaire Est - Hopital Saint-Antoine, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Local Institution - 497, Pierre-Bénite
  - CHU La Miletrie, Poitiers
  - Local Institution - 516, Poitiers
  - CHRU Rennes, Rennes
  - Local Institution - 504, Rennes
  - Institut Universitaire du Cancer de Toulouse (IUCT) - Oncopole, Toulouse
  - CHRU Hopital Bretonneau, Tours
  - Local Institution - 468, Tours
- Germany (12):
  - ChariteUniversitatsmedizinCampus Benjamin Franklin, Berlin
  - Local Institution - 442, Berlin
  - Local Institution - 417, Dresden
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Local Institution - 475, Essen
  - Universitaetsklinikum EssenInnere Klinik und Poliklinik, Essen
  - Local Institution - 496, Freiburg im Breisgau
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Local Institution - 430, Heidelberg
  - University of Heidelberg, Heidelberg
  - Local Institution - 410, Tübingen
  - UKT Universitaetsklinikum Tuebingen, Tübingen
- Greece (8):
  - General Hospital of Athens Evangelismos, Athens
  - Local Institution - 484, Athens
  - Local Institution - 422, Athens
  - University of Athens Medical school - Regional General Hospital, Athens
  - Local Institution - 487, Mezourlo
  - University General Hospital of Larissa, Mezourlo
  - George Papanikolaou General Hospital of Thessaloniki, Thessloniki
  - Local Institution - 465, Thessloniki
- Ireland (6):
  - Local Institution - 462, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Local Institution - 431, Dublin
  - St James Hospital, Dublin
  - Local Institution - 413, Galway
  - University College Hospital Galway, Galway
- Israel (7):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Local Institution - 457, Jerusalem
  - Local Institution - 433, Kfar Saba
  - Meir Medical Center, Kfar Saba
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center Department of Hematology, Tel Aviv
- Italy (24):
  - Local Institution - 449, Bergamo
  - USC Ematologia, Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Local Institution - 456, Bologna
  - Policlinico S. Orsola - Malpighi, Bologna
  - Local Institution - 415, Catania
  - Ospedale Ferrarotto, Catania
  - Local Institution - 403, Modena
  - University of Modena, Modena
  - IRCCS Policlinico San Matteo, Pavia
  - Local Institution - 451, Pavia
  - Azienda Unita Sanitaria Locale (Ausl) Pescara - Presidio Ospedaliero Di Pescara, Pescara
  - Local Institution - 441, Pescara
  - Azienda Ospedaliera di Reggio Emilia - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Local Institution - 414, Reggio Emilia
  - La Sapienza, University of Rome, Rome
  - Local Institution - 460, Rome
  - A.O.U.S. Giovanni e Ruggi d'Aragona UOC UTIC, Salerno
  - Local Institution - 459, Salerno
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Local Institution - 453, San Giovanni Rotondo
  - Azienda Ospedaliera S Maria di Terni, Terni
  - Local Institution - 402, Terni
  - Azienda Ospedaliera San Giovanni Battista, Torino
  - Local Institution - 401, Torino
- Japan (10):
  - Hitachi General Hospital, Hitachi, Ibaraki
  - Local Institution - 620, Hitachi, Ibaraki
  - Kameda Medical Center, Kamogawa
  - Local Institution - 625, Kamogawa
  - Local Institution - 626, Okayama
  - Okayama Medical Center, Okayama
  - Japan Red Cross Medical Center, Shibuya-ku
  - Local Institution - 623, Shibuya-ku
  - Local Institution - 622, Tachikawa
  - National Hospital Organization Disaster Medical Center, Tachikawa
- Netherlands (5):
  - Local Institution - 514, Groningen
  - Universitair Medisch Centrum Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Erasmus Medical Center, Rotterdam
  - Local Institution - 494, Rotterdam
- Norway (3):
  - Local Institution - 412, Oslo
  - Oslo universitetssykehus, Rikshospitalet, Oslo
  - St Olavs Hospital, Trondheim
- Poland (17):
  - Local Institution - 411, Brzozów
  - Szpital Specjalistyczny w Brzozowie, Brzozów
  - Szpital Uniwersytecki nr 2 im dr. Jana Biziela, Bydgoszcz
  - Local Institution - 407, Chorzów
  - Zespol Szpitali Miejskich, Chorzów
  - Klinika Hematologii Akademii Medycznej w Gdansku, Gdansk
  - Local Institution - 463, Gdansk
  - Local Institution - 440, Krakow
  - Oddzial Kliniczny Kliniki Hematologii, Krakow
  - Kopernik Memorial Hospital, Lodz
  - Local Institution - 418, Lodz
  - Klinika Hematoonkologii i Transplantacji Szpiku, Lublin
  - Local Institution - 439, Lublin
  - Local Institution - 437, Poznan
  - Oddzial Hematologii i Chorob Rozrostowych Ukladu Krwiotworczego, Poznan
  - Centrum Onkologii-Instytut im.Marii Sklodowskiej-Curie, Warsaw
  - Local Institution - 448, Warsaw
- Portugal (12):
  - Hospital de Braga, Braga
  - Local Institution - 450, Braga
  - Instituto Portugues de Oncologia de Lisboa, Francisco Gentil, Lisbon
  - Local Institution - 454, Lisbon
  - Fundacao Champalimaud, Lisbon
  - Local Institution - 473, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Local Institution - 466, Lisbon
  - Local Institution - 464, Porto
  - Instituto Portugues de Oncologia do Porto, Francisco Gentil, Porto
  - Local Institution - 425, Porto
  - Hospital de Santo Antonio- Porto, Porto
- Ad-Vance Medical Research, LLC, Ponce, Puerto Rico
- Russia (7):
  - City Clinical Hospital 52, Moscow
  - Local Institution - 521, Moscow
  - Local Institution - 517, Moscow
  - Moscow State Healthcare Institution City clinical hospital n.a. S.P.Botkin, Moscow
  - Local Institution - 520, Nizhny Novgorod
  - State Budgetary Healthcare Institution of Nizhniy Novgorod Region, Nizhny Novgorod
  - Russian Research Institute of Hematology and Transfusiology of the Federal Biomedical Agency, Saint Petersburg
- Spain (16):
  - Hospital Universitari Germans Trias i Pujol Can Ruti, Badalona (Barcelona)
  - Local Institution - 423, Badalona (Barcelona)
  - Hospital Clinic de Barcelona, Barcelona
  - Local Institution - 424, Barcelona
  - Hospital de Basurto-Osakidetza, Bilbao
  - Hospital 12 de Octubre, Madrid
  - Local Institution - 452, Madrid
  - Hospital Morales Meseguer, Murcia
  - Local Institution - 502, Murcia
  - Complejo Hospitalario De Orense, Ourense
  - Local Institution - 526, Ourense
  - Clinica Universidad de Navarra, Pamplona
  - Local Institution - 434, Pamplona
  - Complejo Hospitalario Nuestra Senora de Valme, Seville
  - Local Institution - 492, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sweden (9):
  - Falu lasarett, Falun
  - Local Institution - 426, Falun
  - Local Institution - 478, Gothenburg
  - Sahlgrenska University Hospital, Gothenburg
  - Local Institution - 429, Luleå
  - Sunderby Sjukhus, Luleå
  - Karolinska University, Stockholm
  - Local Institution - 471, Stockholm
  - Sundsvalls sjukhus- Medicinkliniken, Sundsvall
- Turkey (Türkiye) (20):
  - Ankara University Medical Faculty Cebeci Hospital, Ankara
  - Local Institution - 428, Ankara
  - Gazi Universitesi Tip Fakultesi Hastanesi, Ankara
  - Local Institution - 409, Ankara
  - Ankara Universitesi Tip Fakultesi, Ankara
  - Local Institution - 408, Ankara
  - Local Institution - 488, Antalya
  - Medstar Antalya Hospital, Antalya
  - Eskisehir Osmangazi University, Eskişehir
  - Local Institution - 420, Eskişehir
  - Local Institution - 421, Gaziantep
  - Gaziantep University, Gaziantep
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Local Institution - 445, Istanbul
  - Istanbul University Faculty of Medicine, Istanbul
  - Local Institution - 474, Istanbul
  - Ege University Medical School, Izmir
  - Local Institution - 419, Izmir
  - Karadeniz Teknik Universitesi Tip Fakultesi Farabi Hastanesi, Trabzon
  - Local Institution - 404, Trabzon
- United Kingdom (24):
  - The Royal Bournemouth Hospital, Bournemouth
  - Kent and Canterbury Hospital, Canterbury Kent
  - Local Institution - 479, Canterbury Kent
  - Local Institution - 406, Edinburgh Scotland
  - Western General Hospital, Edinburgh Scotland
  - Local Institution - 490, London
  - University College London Hospitals, London
  - Kings College Hospital, London
  - Local Institution - 461, London
  - Local Institution - 512, Oxford
  - University of Oxford, Oxford
  - Derriford Hospital Plymouth Oncology Centre Clinical Trials Unit, Plymouth
  - Local Institution - 515, Plymouth
  - Local Institution - 500, Sheffield
  - Sheffield Teaching Hospitals NHS Foundation Trust - Royal Hallamshire Hospital, Sheffield
  - Local Institution - 493, Southampton
  - Southampton General Hospital, Southampton
  - University Hospital of North Staffordshire Nhs Trust - City General Hospital, Stoke-on-Trent
  - Local Institution - 405, Swansea
  - Singleton Hospital, Swansea
  - Local Institution - 482, Wolverhampton
  - New Cross Hospital, Wolverhampton
  - Local Institution - 436, Worcester
  - Worcestershire Acute Hospitals NHS Trust, Worcester

REFERENCES:
- [Derived] Richardson PG, Oriol A, Beksac M, Liberati AM, Galli M, Schjesvold F, Lindsay J, Weisel K, White D, Facon T, San Miguel J, Sunami K, O'Gorman P, Sonneveld P, Robak P, Semochkin S, Schey S, Yu X, Doerr T, Bensmaine A, Biyukov T, Peluso T, Zaki M, Anderson K, Dimopoulos M; OPTIMISMM trial investigators. Pomalidomide, bortezomib, and dexamethasone for patients with relapsed or refractory multiple myeloma previously treated with lenalidomide (OPTIMISMM): a randomised, open-label, phase 3 trial. Lancet Oncol. 2019 Jun;20(6):781-794. doi: 10.1016/S1470-2045(19)30152-4. Epub 2019 May 13. PMID 31097405
- [Derived] Richardson PG, Hofmeister CC, Raje NS, Siegel DS, Lonial S, Laubach J, Efebera YA, Vesole DH, Nooka AK, Rosenblatt J, Doss D, Zaki MH, Bensmaine A, Herring J, Li Y, Watkins L, Chen MS, Anderson KC. Pomalidomide, bortezomib and low-dose dexamethasone in lenalidomide-refractory and proteasome inhibitor-exposed myeloma. Leukemia. 2017 Dec;31(12):2695-2701. doi: 10.1038/leu.2017.173. Epub 2017 Jun 2. PMID 28642620
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 548 participants treated
Groups:
- Treatment 1: POM+BTZ+LD-DEX: POM (Pomalidomide)
  * 4 mg/day on Days 1 to 14 of each 21-day treatment cycle BTZ (Bortezomib)
  * For Cycles 1 - 8: 1.3 mg/m2/dose on Days 1, 4, 8, and 11 of a 21-day cycle
  * For Cycles 9 onwards: 1.3 mg/m2/dose on Days 1 and 8 of a 21-day cycle DEX (Dexamethasone)
  * For Cycles 1 to 8, 20 mg/day (≤ 75 years old) or 10 mg/day (> 75 years old) on Days 1, 2, 4, 5, 8, 9, 11 and 12 of a 21-day cycle.
  * For Cycles 9 and onward, 20 mg/day (≤ 75 years old) or 10 mg/day (> 75 years old) on Days 1, 2, 8, and 9 of a 21-day cycle.
- Treatment 2: BTZ+LD-DEX: BTZ ((Bortezomib)
  * For Cycles 1 - 8: 1.3 mg/m2/dose on Days 1, 4, 8, and 11 of a 21-day cycle
  * For Cycles 9 onwards: 1.3 mg/m2/dose on Days 1 and 8 of a 21-day cycle DEX (Dexamethasone)
  * For Cycles 1 to 8, 20 mg/day (≤ 75 years old) or 10 mg/day (> 75 years old) on Days 1, 2, 4, 5, 8, 9, 11 and 12 of a 21-day cycle.
  * For Cycles 9 and onward, 20 mg/day (≤ 75 years old) or 10 mg/day (> 75 years old) on Days 1, 2, 8, and 9 of a 21-day cycle.
Period: Randomization
Arm/Group | Treatment 1: POM+BTZ+LD-DEX | Treatment 2: BTZ+LD-DEX
Started | 281 | 278
Completed | 278 | 270
Not Completed | 3 | 8
Not completed — Physician Decision | 0 | 1
Not completed — clinical progression | 0 | 1
Not completed — progressive disease | 0 | 2
Not completed — Withdrew informed consent | 0 | 4
Not completed — Death | 1 | 0
Not completed — Randomization error | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Treatment Period
Arm/Group | Treatment 1: POM+BTZ+LD-DEX | Treatment 2: BTZ+LD-DEX
Started | 278 | 270
Completed | 0 | 0
Not Completed | 278 | 270
Not completed — Lost to Follow-up | 0 | 2
Not completed — Progressive Disease | 167 | 165
Not completed — Adverse Event | 39 | 52
Not completed — Withdrawal of Consent | 25 | 22
Not completed — Death | 20 | 9
Not completed — Other Reasons | 27 | 19
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1: POM+BTZ+LD-DEX | Treatment 2: BTZ+LD-DEX | Total
Number analyzed (Participants) | 281 | 278 | 559
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (10.13) | 66.1 (10.16) | 66.0 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 131 | 257
  Male | 155 | 147 | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 31
  Not Hispanic or Latino | 244 | 241 | 485
  Unknown or Not Reported | 20 | 23 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 8 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 13 | 21
  White | 237 | 234 | 471
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival by Independent Response Adjudication Committee (IRAC)
Description: Progression free survival (PFS) will be calculated as the time between the randomization and progressive disease (PD) or death.
  Progressive Disease is defined as an Increase of ≥ 25% from nadir in:
  * Serum M-component and/or (the absolute increase must be ≥ 0.5 g/dL)g
  * Urine M-component and/or (the absolute increase must be ≥ 200 mg/24 hours)
  * In patients without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels, the absolute increase must be > 100 mg/dL.
  * Bone marrow plasma cell percentage, the absolute % must be ≥ 10%h
  * Definite development of new bone lesions or soft tissue plasmacytomas increase in the size of existing bone lesions or soft tissue plasmacytomas. -Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: From randomization to progressive disease or death during the IRAC assessment period, up to approximately 42 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1: POM+BTZ+LD-DEX | Treatment 2: BTZ+LD-DEX
Number analyzed (Participants) | 281 | 278
Months | 11.20 [9.66 to 13.73] | 7.10 [5.88 to 8.48]
Statistical Analysis 1: Comparison: Treatment 1: POM+BTZ+LD-DEX vs Treatment 2: BTZ+LD-DEX; Test type: Superiority; p = 0.001, Based on Cox proportional hazards model; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.49 to 0.77]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is calculated as the time from randomization to death from any cause.
Time Frame: From randomization to date of death, up to approximately 65 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1: POM+BTZ+LD-DEX | Treatment 2: BTZ+LD-DEX
Number analyzed (Participants) | 281 | 278
Months | 35.58 [28.55 to 41.20] | 31.61 [26.05 to 37.16]
Statistical Analysis 1: Comparison: Treatment 1: POM+BTZ+LD-DEX vs Treatment 2: BTZ+LD-DEX; Test type: Superiority; p = 0.571, Log Rank; The p-value is based on a stratified log-rank test with stratification factors as above Cox model; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.77 to 1.15] — Based on Cox proportional hazards model, comparing the hazard functions associated with treatment groups, stratified by age, prior number of anti-myeloma regimens, and beta-2 macroglobulin at Screening

3. Secondary Outcome: Overall Response Rate by Independent Response Adjudication Committee (IRAC)
Description: The ORR together with the relative proportions in each response category (ie, stringent CR [sCR], CR, very good PR [VGPR], PR, SD, and PD) by treatment using the IMWG criteria will be examined.
  Complete Response: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow
  SCR: CR+ Normal FLC ratio and Absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence
  VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine Mprotein level < 100 mg per 24 hours
  PR: ≥ 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hours
  Progressive Disease: Please refer to Primary outcome measure for definition
  SD: Not meeting criteria for CR, VGPR, PR, or progressive disease
Time Frame: From randomization to progressive disease or death during the IRAC assessment period, up to approximately 42 months
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: POM+BTZ+LD-DEX | Treatment 2: BTZ+LD-DEX
Number analyzed (Participants) | 281 | 278
Participants
  Stringent complete response | 9 | 2
  Complete Reponse | 35 | 9
  Very Good Partial Response | 104 | 40
  Partial Response | 83 | 88
  Stable Disease | 32 | 106
  Progressive Disease | 11 | 16
  Not Evaluable | 7 | 17

4. Secondary Outcome: Duration of Response by Independent Response Adjudication Committee (IRAC)
Description: Duration of myeloma response is defined as the duration from the time when the IMWG response criteria are first met for sCR or CR or VGPR or PR until the first date the response criteria are met for PD or until the subject died from any cause, whichever occurs first.
  Complete Response: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow
  SCR: CR+ Normal FLC ratio and Absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence
  VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine Mprotein level < 100 mg per 24 hours
  PR: ≥ 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hours
  Progressive Disease: Please refer to Primary outcome measure for definition
  SD: Not meeting criteria for CR, VGPR, PR, or progressive disease
Time Frame: From randomization to progressive disease or death during the IRAC assessment period, up to approximately 42 months
Population: All randomized participants with a response (sCR or CR or VGPR or PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1: POM+BTZ+LD-DEX | Treatment 2: BTZ+LD-DEX
Number analyzed (Participants) | 231 | 139
Months | 13.70 [10.94 to 18.10] | 10.94 [8.11 to 14.78]
Statistical Analysis 1: Comparison: Treatment 1: POM+BTZ+LD-DEX vs Treatment 2: BTZ+LD-DEX; Test type: Superiority; p = 0.064, Unstratified log-rank test; The p-value is based on an unstratified log-rank test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.56 to 1.02] — Based on Cox proportional hazards model comparing the hazard functions associated with treatment groups

5. Secondary Outcome: Number of Participants With Grade 3-4 Treatment Emergent Adverse Events (TEAE)
Description: Treatment-emergent adverse events (TEAEs) are defined as any AE occurring or worsening on or after the first dose date of the study treatment and within 28 days after the last dose date.
Time Frame: From first dose to 28 days after the last dose (up to approximately 44 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: POM+BTZ+LD-DEX | Treatment 2: BTZ+LD-DEX
Number analyzed (Participants) | 278 | 270
Participants | 259 | 194

6. Secondary Outcome: Number of Participants With Grade 5 Treatment Emergent Adverse Events (TEAE)
Description: as for outcome 5
Time Frame: From first dose to 28 days after the last dose (up to approximately 44 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: POM+BTZ+LD-DEX | Treatment 2: BTZ+LD-DEX
Number analyzed (Participants) | 278 | 270
Participants | 29 | 12

ADVERSE EVENTS:
Time Frame: AEs and SAEs: From first treatment to 28 days after last dose, up to approximately 44 months on average of 10 months. All-Cause mortality: from randomization to end of the study, approximately 65 months.
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants.
  The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Treatment 1: POM + BTZ + LD-DEX: POM (Pomalidomide)
  * 4 mg/day on Days 1 to 14 of each 21-day treatment cycle BTZ (Bortezomib)
  * For Cycles 1 - 8: 1.3 mg/m2/dose on Days 1, 4, 8, and 11 of a 21-day cycle
  * For Cycles 9 onwards: 1.3 mg/m2/dose on Days 1 and 8 of a 21-day cycle DEX (Dexamethasone)
  * For Cycles 1 to 8, 20 mg/day (≤ 75 years old) or 10 mg/day (> 75 years old) on Days 1, 2, 4, 5, 8, 9, 11 and 12 of a 21-day cycle.
  * For Cycles 9 and onward, 20 mg/day (≤ 75 years old) or 10 mg/day (> 75 years old) on Days 1, 2, 8, and 9 of a 21-day cycle.
- Treatment 2: BTZ + LD-DEX: BTZ ((Bortezomib)
  * For Cycles 1 - 8: 1.3 mg/m2/dose on Days 1, 4, 8, and 11 of a 21-day cycle
  * For Cycles 9 onwards: 1.3 mg/m2/dose on Days 1 and 8 of a 21-day cycle DEX (Dexamethasone)
  * For Cycles 1 to 8, 20 mg/day (≤ 75 years old) or 10 mg/day (> 75 years old) on Days 1, 2, 4, 5, 8, 9, 11 and 12 of a 21-day cycle.
  * For Cycles 9 and onward, 20 mg/day (≤ 75 years old) or 10 mg/day (> 75 years old) on Days 1, 2, 8, and 9 of a 21-day cycle.
Arm/Group | Treatment 1: POM + BTZ + LD-DEX | Treatment 2: BTZ + LD-DEX
All-Cause Mortality (participants affected / at risk) | 197/281 | 193/278
Serious Adverse Events (participants affected / at risk) | 177/278 | 119/270
Other Adverse Events (participants affected / at risk) | 276/278 | 260/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1: POM + BTZ + LD-DEX (N=278) | Treatment 2: BTZ + LD-DEX (N=270)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 1
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 9 | 2
Atrial flutter (Cardiac disorders) | 2 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 3 | 2
Cardiac failure congestive (Cardiac disorders) | 3 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric volvulus (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Death (General disorders) | 4 | 0
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 5 | 9
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 2
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 12 | 5
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Acute hepatitis B (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 2
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchitis pneumococcal (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 4 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Enterobacter pneumonia (Infections and infestations) | 1 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 2 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 2 | 0
H1N1 influenza (Infections and infestations) | 1 | 1
Haemophilus infection (Infections and infestations) | 0 | 1
Herpes oesophagitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 10 | 4
Leishmaniasis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 10 | 5
Lung infection (Infections and infestations) | 2 | 2
Mastoiditis (Infections and infestations) | 0 | 1
Meningitis listeria (Infections and infestations) | 1 | 0
Meningococcal infection (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 34 | 17
Pneumonia bacterial (Infections and infestations) | 2 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 2 | 0
Pneumonia legionella (Infections and infestations) | 2 | 0
Pneumonia moraxella (Infections and infestations) | 1 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 2
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 2 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 2
Pulmonary sepsis (Infections and infestations) | 2 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 5 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 1
Septic shock (Infections and infestations) | 6 | 0
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 3 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 3
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Chest X-ray abnormal (Investigations) | 0 | 1
Coronavirus test positive (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteorrhagia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Scrotal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1
Spinal cord compression (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 6 | 5
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 8 | 6
Anuria (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 4
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1: POM + BTZ + LD-DEX (N=278) | Treatment 2: BTZ + LD-DEX (N=270)
Anaemia (Blood and lymphatic system disorders) | 87 | 72
Leukopenia (Blood and lymphatic system disorders) | 37 | 9
Lymphopenia (Blood and lymphatic system disorders) | 14 | 9
Neutropenia (Blood and lymphatic system disorders) | 150 | 29
Thrombocytopenia (Blood and lymphatic system disorders) | 110 | 105
Atrial fibrillation (Cardiac disorders) | 26 | 5
Cataract (Eye disorders) | 22 | 3
Vision blurred (Eye disorders) | 14 | 9
Abdominal distension (Gastrointestinal disorders) | 17 | 6
Abdominal pain (Gastrointestinal disorders) | 30 | 19
Abdominal pain upper (Gastrointestinal disorders) | 23 | 16
Constipation (Gastrointestinal disorders) | 106 | 65
Diarrhoea (Gastrointestinal disorders) | 102 | 82
Dry mouth (Gastrointestinal disorders) | 19 | 11
Dyspepsia (Gastrointestinal disorders) | 22 | 25
Nausea (Gastrointestinal disorders) | 52 | 56
Stomatitis (Gastrointestinal disorders) | 17 | 1
Vomiting (Gastrointestinal disorders) | 35 | 27
Asthenia (General disorders) | 52 | 48
Fatigue (General disorders) | 107 | 72
Influenza like illness (General disorders) | 15 | 9
Oedema peripheral (General disorders) | 101 | 54
Pyrexia (General disorders) | 72 | 33
Bronchitis (Infections and infestations) | 43 | 20
Conjunctivitis (Infections and infestations) | 26 | 16
Influenza (Infections and infestations) | 27 | 13
Lower respiratory tract infection (Infections and infestations) | 17 | 8
Pneumonia (Infections and infestations) | 26 | 21
Respiratory tract infection (Infections and infestations) | 21 | 16
Upper respiratory tract infection (Infections and infestations) | 71 | 51
Urinary tract infection (Infections and infestations) | 36 | 28
Viral upper respiratory tract infection (Infections and infestations) | 36 | 18
Accidental overdose (Injury, poisoning and procedural complications) | 35 | 11
Fall (Injury, poisoning and procedural complications) | 20 | 11
Alanine aminotransferase increased (Investigations) | 14 | 3
Weight decreased (Investigations) | 20 | 18
Weight increased (Investigations) | 19 | 19
Decreased appetite (Metabolism and nutrition disorders) | 29 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 43 | 28
Hypocalcaemia (Metabolism and nutrition disorders) | 20 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 45 | 31
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 20 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 61 | 38
Bone pain (Musculoskeletal and connective tissue disorders) | 25 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 30 | 16
Muscular weakness (Musculoskeletal and connective tissue disorders) | 41 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 | 38
Dizziness (Nervous system disorders) | 49 | 29
Dysgeusia (Nervous system disorders) | 18 | 8
Headache (Nervous system disorders) | 35 | 25
Hypoaesthesia (Nervous system disorders) | 7 | 15
Paraesthesia (Nervous system disorders) | 18 | 5
Peripheral sensorimotor neuropathy (Nervous system disorders) | 18 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 134 | 103
Syncope (Nervous system disorders) | 14 | 6
Tremor (Nervous system disorders) | 32 | 8
Anxiety (Psychiatric disorders) | 13 | 17
Depression (Psychiatric disorders) | 16 | 7
Insomnia (Psychiatric disorders) | 49 | 54
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 45
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62 | 32
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 16
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Rash (Skin and subcutaneous tissue disorders) | 31 | 11
Hypertension (Vascular disorders) | 24 | 22
Hypotension (Vascular disorders) | 26 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT01734928/Prot_SAP_000.pdf